CLINICAL TRIAL: NCT04629703
Title: Double-Blind, Randomized, Placebo-Controlled, Multi-Center Phase 3 Study to Evaluate the Efficacy and Safety of Fostamatinib in COVID-19 Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-935788-061
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Covid19; SARS (Severe Acute Respiratory Syndrome); SARS Pneumonia; SARS-Associated Coronavirus as Cause of Disease Classified Elsewhere; Pneumonia; Pneumonia, Viral
Keywords: COVID19; SARS-Associated Coronavirus Pneumonia; Pneumonia, Viral
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Pneumonia; Pneumonia, Viral | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fostamatinib (150 mg twice daily for 14 days) + Standard of Care (Active Comparator): Fostamatinib (150 mg twice daily for 14 days) + Standard of Care
  Interventions: Drug: Fostamatinib
- Placebo (twice daily for 14 days) + Standard of Care (Placebo Comparator): Placebo (twice daily for 14 days) + Standard of Care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib (150 mg twice daily) for 14 days and Standard of Care
  Other Names: Fostamatinib disodium
  Arms: Fostamatinib (150 mg twice daily for 14 days) + Standard of Care
Drug: Placebo — Placebo (twice daily) for 14 days and Standard of Care
  Arms: Placebo (twice daily for 14 days) + Standard of Care

SUMMARY:
The study is a double-blind, randomized, placebo-controlled, multi-center, Phase 3 study to evaluate the efficacy and safety of fostamatinib in COVID-19 subjects.

DETAILED DESCRIPTION:
The primary objective of this study is:

To evaluate the efficacy of fostamatinib when used in combination with standard of care (SOC) in subjects hospitalized with COVID- 19 and requiring oxygen supplementation, as measured by days on oxygen.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at screening.
* The subject or a legally authorized representative has provided written informed consent.
* Hospitalized COVID-19 subjects without respiratory failure who are either not receiving any oxygen therapy or are receiving supplemental oxygen via mask or nasal prongs.
* Male or non-pregnant, non-lactating female subjects with SARS-CoV-2 infection documented by a hospital approved diagnostic test (eg, a Food and Drug Administration authorized test in the US) within 7 days prior to randomization.

Exclusion Criteria:

* Pregnant or lactating female of childbearing potential.
* Use of extracorporeal membrane oxygenation (ECMO).
* Uncontrolled hypertension (systolic blood pressure [BP] ≥160 mmHg and/or diastolic BP ≥100 mmHg), unstable angina, congestive heart failure of New York Heart Association classification III or IV, serious cardiac arrhythmia requiring treatment at screening.
* History of myocardial infarction within 1 month prior to screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Number of days on oxygen from randomization on Day 1 to Day 29 | 29 days
  Number of days on oxygen from randomization on Day 1 to Day 29

SECONDARY OUTCOMES:
Mean change from baseline over time in clinical status score using the 8-point ordinal scale, to the average from Day 5 through Day 15. | 10 days
  Mean change from baseline over time in clinical status score using the 8-point ordinal
Number of days in the ICU from randomization on Day 1 to Day 29 | 29 days
  Number of days in the ICU from randomization on Day 1 to Day 29
Time to first sustained hospital discharge by Day 29. (A discharge is defined as sustained when no readmission occurs by Day 29 after the discharge). | 29 days
  Time to first sustained hospital discharge by Day 29. (A discharge is defined as sustained when no readmission occurs by Day 29 after the discharge).
All-cause mortality by Day 29. | 29 days
  All-cause mortality by Day 29.
All-cause mortality by Day 60 | 60 days
  All-cause mortality by Day 60
Proportion of subjects alive by Day 29 and oxygen free on Day 29. | 29 days
  Proportion of subjects alive by Day 29 and oxygen free on Day 29.
Proportion of subjects alive by Day 60 and oxygen free on Day 29 | 60 days
  Proportion of subjects alive by Day 60 and oxygen free on Day 29

CONTACTS AND LOCATIONS:
Locations (46):
- United States (9):
  - University of California Irvine, Orange, California
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Alternative Research Associates, LLC, Hialeah, Florida
  - Alternative Research Associates, LLC, Miami, Florida
  - Loyola University Medical School, Maywood, Illinois
  - Harvard Medical School- Bringham and Women's Hospital, Boston, Massachusetts
  - Henry Ford, Detroit, Michigan
  - Ascension Medical Group- St. John Clinic Infectious Disease, Tulsa, Oklahoma
  - Houston Methodist Research Institute, Houston, Texas
- Argentina (13):
  - Corporacion Medica de General San Martin, San Martín, Buenos Aires
  - Clinica Chutro, Córdoba, CP
  - Hospital Lencinas, Godoy Cruz, Mendoza Province
  - Hospital de Alta Complejidad Cuenta Alta, Buenos Aires
  - Hospital Del Bicentenario - Dr. Luis Federico Leloir, Buenos Aires
  - Clinica Zabala, Buenos Aires
  - Clinica Adventista Belgrano, Buenos Aires
  - Clinica Monte Grande, Buenos Aires
  - Hospital de Infecciosas Dr.Francisco Javier Muñiz, Buenos Aires
  - Sanatorio Guemes, Buenos Aires
  - Sanatorio Sagrado Corazon, Buenos Aires
  - Hospital San Roque, Córdoba
  - Sanatorio Mayo Privado, Córdoba
- Brazil (13):
  - Hospital das Clínicas da Universidade Federal de Goiás (HC/UFG), Goiânia, Goiás
  - Hospital Luxenburgo-Associação Mário Penna, Belo Horizonte, Minas Gerais
  - Hosp. Angelina Caron, Campina Grande do Sul, Paraná
  - Hospital Universitario de Maringa, Maringá, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre - ISCMPA, Porto Alegre, Rio Grande do Sul
  - Hospital des clinicas de porto alegre - Centro de pequisas clinicas, Porto Alegre, Rio Grande do Sul
  - Complexo de Prevenção, Diagnóstico, Terapia e Reabilitação Respiratória LTDA, Blumenau, Santa Catarina
  - Hospital Alemão Oswaldo Cruz (HAOC), Bela Vista, São Paulo
  - Hospital Universitário São Francisco na Providência de Deus, Bragança Paulista, São Paulo
  - Pontificia Universidade Catolica de Campinas (PUC-CAMP) - Hospital e Maternidade Celso Pierro (HMCP), Campinas, São Paulo
  - Hospital Bandeirantes (LeForte), Liberdade, São Paulo
  - Fundação Faculdade Reg. de Med de SJRP, São José do Rio Preto, São Paulo
  - Clinica de Alergia Martti Antila S/S Ltda, Sorocaba, São Paulo
- Mexico (11):
  - Unidad Medica para la Salud Integral (UMSI), Monterrey, Nuevo León
  - Star Medica Vivo Bicentenario, Nezahualcóyotl, State of Mexico
  - Köhler & Milstein Research, Mérida, Yucatán
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Icaro Investigaciones en Medicina, Chihuahua City
  - Nuevo Hospital Civil de Guadalajara, Guadalajara
  - Centro Medico Issemym Toluca, Metepec
  - The American British Cowdray Medical Center I.A.P., Mexico City
  - Hospital Ángeles Roma, México
  - CEPREP Centro de Prevención y Rehabilitación de Enfermedades Pulmonares Crónicas, Nuevo León
  - Hospital Civil de Culiacan, Sinaloa

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343